CLINICAL TRIAL: NCT04647513
Title: Evaluation of the Efficacy and Safety of Three Injectable Hyaluronic Acid-based Fillers: Art Filler® Fine Lines, Art Filler® Universal and Art Filler® Lips
Acronym: AF4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires FILLMED (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF4:2018-A02466-49
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Loss of Face Volume
MeSH Terms: interventions — Injections, Intradermal

STUDY DESIGN:
Intervention Model Description: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips). To this end, subjects in whom a correction of at least one of the studied zones is sought, will be included. The aesthetic correction will be appreciated at 3 weeks. Subjects will be followed over 18 months. The persistence of the correction will be evaluated at 3, 6, 9, 12, 15 and 18 months.
  Around 200 subjects aged more than 19 years old with following distribution:
  * Art Filler Fine Lines
  * Forehead wrinkles
  * Upper lip wrinkles
  * Cheek folds
  * Crow's feet wrinkles
  * Art Filler Universal
  * Volume of the lips (for soft volumizing effect)
  * Nasolabial folds alone or with marionette lines
  * Art Filler Lips
  * Volume of the lips (for plumped lips)
  * Very deep Nasolabial folds alone or with marionette lines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Art Filler Fine Lines (forehead) (Experimental): Injection of Art Filler Fine Lines in Forehead wrinkles
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Fine Lines (upper lip) (Experimental): Injection of Art Filler Fine Lines in upper lip wrinkles
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Fine Lines (cheek folds) (Experimental): Injection of Art Filler Fine Lines in cheek folds
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Fine Lines (crow's feet) (Experimental): Injection of Art Filler Fine Lines in crow's feet
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Universal (lips volume) (Experimental): Injection of Art Filler Universal in lips
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Universal (nasolabial folds) (Experimental): Injection of Art Filler Universal in nasolabial folds
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Lips (lips volume) (Experimental): Injection of Art Filler Lips in lips
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)
- Art Filler Lips (very deep nasolabial folds) (Experimental): Injection of Art Filler Lips in very deep nasolabial folds
  Interventions: Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips)

INTERVENTIONS:
Device: Intradermal injection (superficial dermis for Art Filler Fine Lines / moderately deep to deep dermis for Art Filler Universal and Art Filler Lips) — The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume and the aging process. These fillers (also known as soft tissue augmentation medical devices) can correct the skin depressions/wrinkles, balance the disproportions or correct topographical anomalies.

SUMMARY:
The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume and the aging process. These fillers (also known as soft tissue augmentation medical devices) can correct the skin depressions/wrinkles, balance the disproportions or correct topographical anomalies.

In this context, it is proposed to carry out in post-CE marking, an open, prospective and non-comparative study in order to document an adequate aesthetic correction of the most frequent areas treated with Art Filler Fine Lines, Art Filler Universal and Art Filler Lips as well as their immediate and long-term tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who had signed a written informed consent
2. Man or Woman aged ≥ 19 years old
3. Subject having a Fitzpatrick Phototype I to IV
4. Subject having a score of ≥ 1 in the Global aesthetic scale scoring system on at least one area of interest (forehead wrinkles, upper lip wrinkles, cheek folds, crow's feet wrinkles, nasolabial folds and/or marionette wrinkles) and/or ≤ 2 for the lip volume
5. Subject having at least one of the following scales by clinical scoring

   * For subjects injected by Art Filler Fine Lines:
   * a grade ≥ 3 and ≤ 6 on the upper lip wrinkles scale from Bazin
   * a grade ≥ 3 and ≤ 5 on the cheek folds scale from Bazin
   * For women :
   * a grade ≥ 2 and ≤ 5 on the forehead wrinkles scale from Bazin
   * a grade ≥ 2 and ≤ 6 on the crow's feet wrinkles scale from Bazin
   * For men :
   * a grade ≥ 2 and ≤ 6 on the forehead wrinkles from Bazin
   * a grade ≥ 2 and ≤ 6 on the crow's feet wrinkles from Bazin
   * For subjects injected by Art Filler Universal:
   * a grade ≥ 0 and ≤ 2 on the lip volume fullness scale from Medicis (if the subject would like a soft effect on his/ her lips)
   * For women, a grade ≥ 2 and ≤ 4 on the nasolabial folds scale from Bazin
   * For men a grade ≥ 2 and ≤ 4 on the nasolabial folds scale from Bazin
   * For subjects injected by Art Filler Lips:
   * a grade ≥ 0 and ≤ 2 on the lip volume fullness scale from Medicis (if the subject would like a plumpled effect on his/ her lips)
   * For women, a grade of 5 on the nasolabial folds scale from Bazin
   * For men a grade ≥ 5 on the nasolabial folds scale from Bazin
6. Subject registered with health insurance regimen
7. Woman agreeing to take a pregnancy test

Exclusion Criteria:

1. Subject currently participating in another clinical study related to pharmaceuticals or medical devices or being in exclusion period of another clinical study.
2. Subject deprived of freedom by an administrative or legal decision
3. Subject who has received indemnification of 4500 € during the 12 previous months for his/her participation in clinical trials (including participation in this study).
4. Subject who had facial injections/implants of any non-absorbable fillers in her/his whole life.
5. Subject who had laser sessions for skin rejuvenation or laser resurfacing during the 12 previous months or a surgical facelift during the 2 years before the study.
6. Subject with a history of facial aesthetic injection (hyaluronic acid within the previous year, botulinum toxin within the last 6 months and long-term temporary injectable implants (semi-permanent implants) within the previous 2 years).
7. Subject with a skin-retaining device on the face (mesh, gold wire, liquid silicone or other particulate material).
8. Subject who underwent a non-invasive rejuvenation method such as moderate to deep peeling, ultrasound, radiofrequency devices or lasers within the last 6 months.
9. Subject with a history of severe multiple allergies or anaphylactic shock.
10. Subject with a known hypersensitivity to hyaluronic acid, Lidocaine and/or other components of Art Filler Fine Lines®, Art Filler Universal® and Art Filler Fine Lips® solutions.
11. Subject with a known hypersensitivity to chlorhexidine.
12. Subject with a known hypersensitivity to lidocaine or local amide anesthetics.
13. Subject tending to develop inflammatory skin diseases or hypertrophic scars.
14. Subject with a history of streptococcal disease (recurring angina, rheumatic fever).
15. Subject with oral or injectable corticoid treatment (or not stopped for at least 3 months). Inhaled corticoids are permitted as well as topical corticotherapy not involving the head or the neck.
16. Subjects with any concomitant treatment (or not stopped for at least a year) by immunosuppressant or chemotherapy.
17. Subject with a history of radiotherapy involving the head and the neck within the previous year.
18. Subject with a history or a disease associated to the autoimmune or connective tissue disease.
19. Subject presenting on his/her face any skin disease, or an acute inflammatory reaction or a bacterial/viral infection or who had such an episode within the previous 6 weeks.
20. Subject who took aspirin or anticoagulants at regular doses in the last 15 days prior to the act.
21. Subject who has permanently been exposed to the sun or the UV during the last 15 days.
22. Subject with a general pathology, skin disease, dermatosis, acute or chronic systemic disease, and/or taking a general or topical treatment that in the opinion of the investigator may interfere with the treatment or compromise the subject's participation in the study
23. Pregnant or lactating woman.
24. Subject with epilepsy not controlled by treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Correction on D21 assessed with the global clinical aesthetic score | D21 (21 days after the injections)
  Objectively measure the improvement according to a global Aesthetic clinical scoring from D0 to D21 of
  * after injection of Art Filler Fine lines
    * forehead wrinkles (at least 30 subjects)
    * upper lip wrinkles (at least 30 subjects)
    * cheek folds (at least 30 subjects)
    * crow's feet wrinkles (30 subjects)
  * after injection of Art Filler Universal
    * lips volume (at least 30 subjects)
    * nasolabial folds alone or with marionette wrinkles (at least 30 subjects)
  * after injection of Art Filler Lips
    * lips volume (at least 30 subjects)
    * Very deep nasolabial folds alone or with marionette wrinkles (at least 30 subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Ferial Fanian, MD, Study Director — Laboratoires FILLMED
Locations (1):
- Dr Mihai Gorj, Paris, France

IPD SHARING:
Plan to Share IPD: No